CLINICAL TRIAL: NCT02805036
Title: Comparison of the Hemodynamic Safety of Two Common Alveolar Recruitment Manoeuvres With Regard to Cardiac Output in a Surgical Intensive Care Unit: a Randomized Study
Brief Title: Comparison of the Hemodynamic Safety of Two Common Alveolar Recruitment Manoeuvres With Regard to Cardiac Output in a Surgical Intensive Care Unit
Acronym: RHERA1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0002
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Positive-Pressure Respiration
Keywords: alveolar recruitment; stroke volume/physiology; cardiac output/physiology
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 30 cmH20 for 30 seconds: plateau pressure is hold on at 30 cmH20 pour 30 seconds. The cardiac output and the lung aeration is assessed by ultrasound measures at 3 times: before, at the end of the recruitment and 30 minutes later.
  echocardiography - arterial oximetry
  Interventions: Device: echocardiography; Device: Arterial oximetry
- 10 cmH20 above: plateau pressure is hold on at 10 cmH20 above. The cardiac output and the lung aeration is assessed by ultrasound measures at 3 times: before, at the end of the recruitment and 30 minutes later.
  echocardiography - arterial oximetry
  Interventions: Device: echocardiography; Device: Arterial oximetry

INTERVENTIONS:
Device: echocardiography — • Prospective, simultaneous recording of the cardiac output (measured non-invasively via transthoracic echocardiography) and a number of parameters commonly monitored in the surgical intensive care unit (CVP, SBP/DBP/MBP).
Device: Arterial oximetry — measured by co-oximetry of a blood sample taken via the arterial catheter implemented for critical care

SUMMARY:
Protective ventilation - combining a low tidal volume (between 6 and 8 ml/kg) and alveolar recruitment (AR) manoeuvres repeated every 30 minutes - is currently the standard of care for decreasing morbidity associated with mechanical ventilation.

In contrast, there is no consensus on the type of recruitment manoeuvre, which varies from one centre to another and from one study to another.

The investigators intend to compare two currently used AR techniques with regard to their ventilatory efficacy and hemodynamic safety:

* An end-tidal plateau at 30 cmH20 for 30 seconds.
* An end-tidal plateau at 10 cmH20 above the patient's plateau pressure for 30 seconds, without exceeding 30 cmH20.

ELIGIBILITY:
Inclusion Criteria:

* All sedated, intubated, mechanically ventilated adult patients (over-18) admitted to the surgical intensive care unit and equipped with a central venous catheter and an arterial catheter.
* Good echogenicity
* Social security coverage

Exclusion Criteria:

* Pregnancy
* Cardiac arrhythmia
* Poor echogenicity
* Legal guardianship or incarceration
* Systolic blood pressure ≤90 mmHg
* Respiratory distress
* Patients admitted on an emergency basis (first 24 hours), i.e. not for elective surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sedated, intubated, mechanically ventilated adult patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Variations in cardiac output induced by each type of AR manoeuvre | Day 0

SECONDARY OUTCOMES:
Variations in PaO2 variations induced by each type of AR manoeuvre | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LORNE, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France